CLINICAL TRIAL: NCT04751552
Title: Effect of Erector Spinae Plane Block on Postoperative Pain Intensity in Patients Undergoing Thoracoscopic Surgery: a Randomized Clinical Trial.
Brief Title: Erector Spinae Block for Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Leon Timmerman, MD, PhD, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L20.047
Record Dates: First submitted 2020-10-14; First posted 2021-02-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain; Thoracic Neoplasms
Keywords: Thoracoscopy; Pain; Regional anaesthesia
MeSH Terms: conditions — Pain, Postoperative; Thoracic Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled double blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levobupivacaine group (Active Comparator): Patients receive an ESPB with the local anaesthetic levobupivacaine
  Interventions: Procedure: Erector Spinae Plane Block (for postoperative pain relief)
- Placebo group (Placebo Comparator): Patients receive an ESPB with 0,9% saline
  Interventions: Procedure: Erector Spinae Plane Block (for postoperative pain relief)

INTERVENTIONS:
Procedure: Erector Spinae Plane Block (for postoperative pain relief) — A ultrasound guided single bolus injection of 20 ml of levobupivacaine or placebo between the erector spinae muscle and process transversus of vertebra T5.

SUMMARY:
This randomized clinical trial compares the effects of the erector spinae plane block with levobupivacaine and 0,9% saline on postoperative pain intensity, and opioid consumptions following thoracoscopic pulmonary surgery.

DETAILED DESCRIPTION:
Sixty patients planned for thoracoscopic pulmonary surgery are randomly assigned to an erector spinae plane block (ESPB) with levobupivacaine (intervention group) or 0,9% saline (control group). ESPB is performed under general anaesthesia before surgery.

Postoperative pain medication incudes acetominophen, NSAIDs en parenteral morphine (patient controlled analgesia).

Following surgery pain intensity (numeric rating scale) is registered at the recovery ward one hour after surgery. Furthermore, pain intensity is registered 2,4,8, 12 hours after the operation. On the first postoperative day, pain intensity is registered at 8.00 o'cock AM and 8.00 o'clock PM. Opioid consumption is registered as a second parameter of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracoscopic pulmonary sleeve resection or lobectomy
* Age 18 years or older

  * American Society of Anesthesiologists (ASA) health status class I-III
  * Informed consent

Exclusion Criteria:

* Contraindication for regional analgesia (e.g. coagulopathy, infection at injection site)
* Contraindication for NSAIDs
* Chronic opioid use
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity (numeric rating scale (NRS) (0=no pain up to 10=most pain imaginable) 2 hours after surgery. | 2 hours postoperatively
  Pain level 2 hours after surgery
Pain intensity (NRS) 4 hours after surgery. | 4 hours postoperatively
  Pain level 4 hours after surgery
Pain intensity (NRS) 8 hours after surgery. | 8 hours postoperatively
  Pain level 8 hours after surgery
Pain intensity (NRS) 12 hours after surgery. | 12 hours postoperatively
  Pain level twelve hours after surgery

SECONDARY OUTCOMES:
Pain intensity (NRS) at 8.00 o'clock on the first postoperative day | At 8 o'clock AM on the first postoperative day
  Pain level at 8.00 o'clock on the first postoperative day
Pain intensity (NRS) at 20.00 o'clock on the first postoperative day | At 8 o'clock PM on the first postoperative day
  Pain level at 20.00 o'clock on the first postoperative day
Opioid consumption | First 48 hours after surgery, recorded following disconnection of the PCA device at 8 o'clock AM on the second postoperative day.
  Parenteral morphine use (mg) as recorded by the Patient-Controlled Analgesia (PCA) device
length of stay in recovery ward (minutes) | First 48 hours after surgery
  length of stay in recovery ward (minutes) after surgery
Patient satisfaction of pain therapy | Measurement in the morning of the second postoperative day
  Patient satisfaction of pain therapy (numeric rating scale 0-10(0=severely dissatisfied up to 10= maximally satisfied)
Presence of side effects | First 48 hours
  Daily scoring of side effects (nausea, drowsiness, pruritus, other (yes/no))

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Relevant participant data underlying the final results and conclusions of the study.
Supporting Information: Study Protocol
Time Frame: Following the report of the study